CLINICAL TRIAL: NCT01871298
Title: Exploratory Study of Drug User Health-related Internet and Mobile Technology Use
Brief Title: Drug User Internet and Mobile Tech Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Silvia Cunto-Amesty, Assistant Professor, Columbia University
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: AAAL6402; 1R21DA034841-01A1 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Drug Abuse Illicit
Keywords: internet and mobile technology use; history of drug use; injection drug user (IDU) syringe customers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Website access (Other): While this pilot intervention is not a randomized trial, study participants who report internet use at least once a month will told of a Pilot Website Evaluation Component that they will be able to access for a 4-week study period. This website will contain a educational information tailored to the health needs of drug users. Web content will be similar to materials and public health messages released by the NYC Department of Health and therefore, harm is not likely to arise from viewing such content.
  Interventions: Other: Pilot Website Evaluation Component
- No website access (No Intervention): Participants who report internet use less than once a month will not receive access to the Pilot Website Evaluation Component.

INTERVENTIONS:
Other: Pilot Website Evaluation Component — The pilot health website will contain educational health information such as: health-related videos, searchable map of HIV prevention and other needed health and social services, and the option to register for automatic text message updates on relevant health information.
  Arms: Website access

SUMMARY:
The purpose of this exploratory study is to examine factors associated with frequency and type of internet and mobile technology use among illegal drug users, specifically use of internet and text-messaging to obtain health care information and engage in health care utilization, specifically human immunodeficiency virus (HIV) prevention and treatment services. We will target high drug activity neighborhoods in New York City and enroll participants recruited through targeted street outreach. All participants (n=336) will undergo an audio computer-assisted self-interview (ACASI) that will assess sociodemographics, health care access and utilization, sex/drug use behavior, health status, and characteristics of general and health-related internet/mobile technology use including factors that promote or hinder use. Participants identified as using the internet ≥1/month (n=151) will return for a 4-week ACASI to report on use of the pilot website (which will largely display information currently available in the community in print/ pamphlet/ video form).

DETAILED DESCRIPTION:
At the enrollment visit participants deemed eligible after screening will be consented, and given a 30 minute baseline ACASI survey. At the end of the baseline visit, those participants who reported internet use at least 1x/month (in the past month) will be offered participation in the Pilot Website Evaluation Component. For this component, participants will be instructed on how to use an educational website with health resources. Their use of the website will be tracked. They will be given an appointment to return in 4-weeks for a follow up survey at the pharmacy and a 2-week locator call.

ELIGIBILITY:
Inclusion Criteria:

* any lifetime illegal drug use
* age > 18

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percent of participants who use the pilot website | 4 weeks

SECONDARY OUTCOMES:
Percent of participants who use the internet | Baseline
Percent of participants who use the internet at least once a month | Baseline
Percent of participants who use the internet for health-related purposes | Baseline
Percent of participants who are willing to use internet or mobile technology for health-related purposes | Baseline
Percent of participants who sign up for receipt of automatic text message updates on relevant health information | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Cunto-Amnesty, MD, Principal Investigator — Assistant Professor of Medicine and Population and Family Health, Dept of Medicine Family Med
Locations (1):
- Columbia University Medical Center, New York, New York, United States